CLINICAL TRIAL: NCT01897467
Title: Effect of a Wii Fit Intervention on Balance, Muscular Fitness, and Bone Health in Middle-aged Women
Brief Title: Effect of a Wii Fit Intervention on Components of Fall Risk in Middle-aged Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WiiFit
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Falls; Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): The control is a "wait-list" control, and will have the option to participate in the intervention at the end of the initial 12-week study period. The control group will be asked to not change any of their dietary or exercise habits over the course of the 12 weeks.
  Interventions: Behavioral: Wait-List Control
- Wii Fit (Experimental): Participants in the intervention group will be assigned a Wii console and a Wii Fit balance board. The intervention group will be asked to play for 30 minutes a day, 3 times per week, using only the participant profile pre-programmed for them. They will complete yoga poses and strength training exercises for the first 10 minutes and balance coordination games for the remaining 20 minutes. They will be asked to complete each exercise at least twice, preferably by cycling through all exercises. Participants will be asked to do all of the exercises in one 30-minute session, rather than breaking them up throughout the day.
  All participants will be asked to keep a record of which games they play and for how long. The Wii Fit software also keeps a digital record of which exercises were completed and how long they were performed. At the end of the intervention the investigator will use the information stored in the Wii, as well as activity logs, to assess compliance.
  Interventions: Behavioral: Wii Fit

INTERVENTIONS:
Behavioral: Wii Fit — Exercises to be done on the Wii Fit include: warrior pose, half-moon pose, lunges, side lunges, balance bubble, ski slalom, soccer heading, and table tilt.
  Other Names: Nintendo Wii Fit Intervention
  Arms: Wii Fit
Behavioral: Wait-List Control — Participants maintain currently physical activity and diet habits for 12 weeks. They have the option to participate in the intervention at the end of the 12-week period, but it is not mandatory.
  Arms: Control

SUMMARY:
Losses of muscular fitness/balance are common occurrences with aging that can lead to an increased fall-risk. The accelerated bone loss that may accompany menopause makes some women even more "at-risk" for serious consequences related to falling. Interventions to reduce fall-risk have been conducted in an attempt to improve balance or muscular fitness, but often these interventions require monotonous exercises that don't arouse enough long-term interest to elicit the improvements. In other words, while the intervention may be beneficial, participants quit before they can realize any gains.

Currently, there is little research that uses novel technology-based programs to promote balance exercises among middle-aged women. The Wii Fit system includes various strength and balance exercises integrated into games intended to have the participant have fun and retain interest, while also improving fitness. By using such a program, women could potentially improve their balance and decrease their fall risk in a way that is fun and exciting.

The purpose of this study is to investigate the effect of a Wii Fit based exercise program on balance/muscular fitness/markers of bone health in women between the ages of 45-60 with low bone mass. Volunteers who have moderately low bone levels (n = 28) will be randomly assigned to either the Wii Fit exercise intervention or a normally active control. Balance ability, muscular fitness, body composition, physical activity levels and markers of bone health will be assessed before and after the intervention.

Each participant in the intervention will be provided a pre-programmed Wii Fit console and balance board to use at home. The intervention will consist of a 12-week program that they perform 30 minutes a day 3 days a week. The exercises include 10 minutes of Yoga poses and strength exercises and then 20 minutes of balance games such as soccer heading, ski slalom and table tilt.

At the 6 week point and the conclusion of the intervention, participants will come to the lab for testing on the same tests done initially.

The overall goal of this study is to gauge the efficacy of this intervention to improve balance, fitness, and bone health in at-risk women. This project is important because it offers an exciting, fun, and motivating way to impact fall-risk before clinical symptoms develop. Overall, this intervention could significantly reduce healthcare dollars spent on fall-related outcomes, as well as reduce fall-related mortality.

ELIGIBILITY:
Inclusion Criteria:

* apparently healthy women between the ages of 45-60
* no contraindications to walking or standing
* no hormonal replacement therapy or any medications or supplements (except for calcium, vitamin D, multivitamin) that affect the bone
* Any vitamin supplements must be over-the-counter (OTC) and cannot be prescription grade.

Exclusion Criteria:

* Those who do not pass the PAR-Q+ (contraindicated for exercise)
* DXA t-score greater than 0 (Note: any woman who has a t-score less than -1.5 will be referred to their health care provider for further follow up and will not be allowed in the study with the approval of their health care professional.)

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Balance | 12 weeks
  Balance will be assessed using the Berg Balance Scale and the FICSIT-4 at baseline, 6-weeks, and 12-weeks.

SECONDARY OUTCOMES:
Muscular Fitness | 12 weeks
  Muscular strength and endurance will be assessed using an isokinetic dynamometer. The strength protocol will involve 60 degrees/second, 180 degrees/second, and 240 degrees/second. Muscular endurance will be assessed via 50 repetitions at 240 degrees/second. Testing will occur at baseline, 6 weeks, and 12 weeks.
Bone Turnover | 12 weeks
  Biomarkers of bone turnover (osteocalcin and c-telopeptide) will be assessed via venous blood draw at baseline, 6 weeks, and 12 weeks.

OTHER OUTCOMES:
Body Composition | 12 weeks
  Total lean mass and fat mass will be assessed via dual-energy x-ray absorptiometry at baseline and 12 weeks.
Bone Mineral Density | 12 weeks
  Bone mineral density (total body) will be assessed via dual-energy x-ray absorptiometry at baseline and 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah J Wherry, MS, Principal Investigator — Arizona State University; Pamela D Swan, PhD, Study Chair — Arizona State University
Locations (1):
- Arizona Biomedical Collaborative, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Wherry SJ, Ananian C, Swan PD. Feasibility of a Home-Based Balance Intervention in Middle-Aged Women Using Wii Fit Plus(R). J Phys Act Health. 2019 Sep 1;16(9):736-744. doi: 10.1123/jpah.2018-0265. Epub 2019 Jul 17. PMID 31310993